CLINICAL TRIAL: NCT04764006
Title: A Single Arm, Open-label, Single Center Phase II Study of Surufatinib Combined With PD-1 in Patients With Advanced MSS-Type Colorectal Cancer Treated With Standard First-line Therapy
Brief Title: Surufatinib Combined With Sintilimab for Advanced MSS-Type Colorectal Cancer : a Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-C101
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-02

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib plus Sintilimab (Experimental): Drug: Surufatinib plus Sintilimab Surufatinib will be given orally. Sintilimab will be given intravenously
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib(250mg ,qd,po)+Sintilimab(200mg,q3w,iv),21 days for a cycle.The curative effect was evaluated every 8 weeks.
  Other Names: HMPL-012

SUMMARY:
A phase II study to assess the efficacy and safety of Surufatinib combined with Sintilimab as a second-line treatment in patients with advanced MSS-Type CRC.

ELIGIBILITY:
Inclusion Criteria:

1. For inclusion in study, patient must provide a written informed consent.
2. Male or female, age18-75 years.
3. Pathologically confirmed unresectable locally advanced or advanced MSS-Type metastatic colorectal adenocarcinoma .
4. The patient had previously failed standard first-line systemic chemotherapy,Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if 6 months or more have passed since completion of therapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
6. Life expectancy > 12 weeks.
7. Have measurable disease based on RECIST 1.1.

Exclusion Criteria:

1. Any therapy with anti-PD-1, or anti-PD-L1/l2 antibodies or anti-cytotoxic T lymphocyte associated antigen-4 (CTLA-4) antibody (or any other antibody acting on T cell costimulatory or checkpoint pathway) or fruquintinib treatment in previous.
2. Prior receipt of Surufatinib.
3. History of any active autoimmune disease or autoimmune disease, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, pituitary inflammation, vasculitis, systemic lupus erythematosus, etc. (except patients with hypothyroidism that can be controlled only by hormone replacement therapy and patients with type I diabetes who only need insulin replacement therapy).
4. History of gastrointestinal perforation and/or fistula, ileus, inflammatory bowel disease, or extensive enterotomy (partial colectomy or extensive enterotomy with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within 6 months prior to first dosing.
5. Any life-threatening bleeding event or grade 3 or 4 bleeding requiring blood transfusion, endoscopy, or surgery with 3 months prior to dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib Combined With Chemotherapy as second-line therapy to Advanced CRC, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Fujian, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided